CLINICAL TRIAL: NCT01276002
Title: Randomized Multicenter Study on Pancreatic Duct Stenting in Disrupted or Obstructed Ducts in Context With Endoscopic Treatment of Pancreatic Pseudocysts.
Brief Title: Evaluation of Pancreatic Duct Stenting in Patients With Pancreatic Pseudocysts.
Acronym: Disduct
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No appropriate participants
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Head Interdisciplinary Endoscopy, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKSH-122010
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Chronic Acute Pancreatitis
Keywords: disrupted duct; pancreatic pseudocysts
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No stenting (No Intervention): Control group, no stenting of the pancreatic duct in case of a disrupted duct
- Pancreatic duct stenting (Active Comparator): in case of a disrupted pancreatic duct, patients will undergo pancreatic duct stenting in this arm
  Interventions: Procedure: pancreatic duct stenting

INTERVENTIONS:
Procedure: pancreatic duct stenting — in case of a disrupted pancreatic duct, patients will undergo pancreatic duct stenting.
  Arms: Pancreatic duct stenting

SUMMARY:
The disruption of the pancreatic duct seems to be a major cause pseudocyst formation and persistence in patients suffering from acute/chronic pancreatitis. No prospective randomized studies have been conducted on the influence of pancreatic duct stenting for the patients' benefits and recurrence rates. The aim fo this study is therefore to evaluate prospectively in a randomized, controlled fashion in patients wit pancreatic pseudocysts, wether pancreatic duct stenting of a disrupted pancreatic duct is beneficial in terms of quicker clinical recovery and avoidance of recurrence of pancreatic pseudocysts.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic pseudocyst, at least 6 cm in diameter
* symptomatic pancreatic pseudocyst
* increasing size of pancreatic pseudocyst within 6 weeks

Exclusion Criteria:

* Pregnancy
* Age less than 18 years
* Postoperative status preventing access to papilla
* Allergy to contrast preventing from ERP
* Missing informed consent to study
* PTT above 1.5 times of normal, unless substituted
* Platelet count less than 50.000/µl, unless substituted
* Pancreatic ascites or fistula
* Life expectancy less than 2 years
* Percutaneously drained cysts are not part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of pancreatic pseudocyst | two years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ellrichmann, MD, Principal Investigator — Interdisciplinary Endoscopy, University hospital Schleswig-Holstein, Campus Kiel, Germany; Annette Fritscher-Ravens, MD, PhD, Study Director — Interdisciplinary Endoscopy, University hospital Schleswig-Holstein, Campus Kiel, Germany
Locations (1):
- Interdisciplinary Endoscopy, University hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany